CLINICAL TRIAL: NCT03999008
Title: A Multicentre, Prospective, Randomized, Placebo Controlled, Double-blinded Study to Demonstrate Potential and Beneficial Effects of Oral Viscous Budesonide (OVB) in the Prevention of Recurrence of Anastomotic Stricture in Children Operated on for Esophageal Atresia With Recurrent Anastomotic Strictures
Brief Title: Oral Viscous Budesonide in Anastomotic Stricture After Esophageal Atresia Repair (OVB in EA)
Acronym: OVB in EA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Christophe Faure, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OVB in EA
Record Dates: First submitted 2019-06-14; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Atresia; Anastomotic Stenosis
MeSH Terms: conditions — Esophageal Atresia | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide (Active Comparator): Oral viscous budesonide will be given in apple sauce according to body weight at inclusion:
  < 10 kg: 250 mcg BID in 5 ml apple sauce 10 kg to <15 kg: 500 mcg BID in 5 ml apple sauce >15 kg: 1000 mcg BID in 5 ml apple sauce
  Interventions: Drug: Budesonide Oral
- Placebo (Placebo Comparator): Placebo: 5 ml apple sauce BID plus 1 mL saline
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Budesonide Oral — The subjects will be included at time of the first dilation for an anastomotic stricture.
  Basal physical exam and clinical evaluation (weight and height, dysphagia score, gastroesophageal reflux, feeding problems, respiratory symptoms, other symptoms).
  Randomization will be conducted by centre. Because long gap esophageal atresia, high tension anastomosis and history of anastomotic leak are reported as risk factors for occurrence of anastomotic strictures, a stratification at randomization will be performed according to these criteria in each centre.
  OVB or placebo will be given by the parents and started the day of the dilation at the first meal after recovering of the dilation and anesthesia.
  Parents will be asked to bring the empty caps which will be counted for assessment of compliance.
  Arms: Budesonide
Drug: Placebos — Apple Sauce 5 mL+ 1 mL saline
  Arms: Placebo

SUMMARY:
The aim of this study is to perform a multicentre, prospective, randomized, placebo controlled, double-blinded study to demonstrate the potential and beneficial effects of OVB in the prevention of recurrence of anastomotic stricture in children operated for esophageal atresia with an anastomotic stricture.

ELIGIBILITY:
Inclusion Criteria:

* Children aged > 1 month to 3 years
* Operated for an esophageal atresia of all types except pure TEF.
* Presence of an anastomotic stricture defined according to experts recommendations :

  * a relative esophageal narrowing at the level of the anastomosis,
  * demonstrated by a contrast study and/or an endoscopy
  * with significant functional impairment and associated symptoms requiring dilation.
  * Symptoms include: feeding or swallowing difficulties, coughing and choking during feeds, food impaction, regurgitation/vomiting of undigested food, drooling. In very young patients: apnea and food refusal.
* Receiving an ongoing treatment by PPI 1 to 2 mg/kg die
* Informed parental consent

Exclusion Criteria:

* Known immune deficiency
* Acute respiratory or intestinal infection
* Severe respiratory, cardiac or neurological condition precluding OVB or placebo swallowing
* Child fed exclusively via nasogastric tube or gastrostomy
* Absence of parental consent

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
number of dilations needed after randomization (beginning of treatment) | 12 months
  number of dilations needed after randomization (beginning of treatment)

SECONDARY OUTCOMES:
Number of patients needing dilation after randomization (beginning of treatment) | 12 months
  Number of patients needing dilation after randomization (beginning of treatment)
Number of patients needing more than 3 dilations after randomization | 12 months
  Number of patients needing more than 3 dilations after randomization
Mean time to further dilation | 12 months
  Mean time to further dilation
Number of patients treated with an adjuvant therapy | 12 months
  Number of patients treated with an adjuvant therapy
Ability to tolerate normal food for age | 12 months
  Ability to tolerate normal food for age
Dysphagia score | 12 months
  Dysphagia score
Quantification of the anastomostic stricture by the Stricture index (SI) calculated on barium swallow at 12 months of age | 12 months
  Quantification of the anastomostic stricture by the Stricture index (SI) calculated on barium swallow at 12 months of age
Side effects/Adverse events | 12 months
  Side effects/Adverse events

IPD SHARING:
Plan to Share IPD: No